CLINICAL TRIAL: NCT01942798
Title: Evaluation of the WiiFit to Enhance Walking in Older Adults With Lower Limb Amputation
Brief Title: Study of WiiFit to Enhance Walking in Older Adult Amputees
Acronym: WiiNWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H13-01858
Record Dates: First submitted 2013-08-27; First posted 2013-09-16 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lower Limb Amputation; Older Adults
Keywords: Rehabilitation; Lower Limb Amputation; Prosthetic; Walking; unilateral transtibial amputation; unilateral transfemoral amputation; older adults; cognitive computer games; home-based training; Nintendo Wii; virtual reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Games (Active Comparator): The Cognitive Games group will receive 40 minute supervised group training three times per week for a period of four weeks. The group for the first week will be held at the clinic, while the remaining three weeks be conducted at the subject's home and supervised by the Trainer remotely using a tablet with video conferencing capability. At the end of the four-week Supervised Phase, subjects will retain the Wii units and they will be encouraged to use the program on their own for an additional period of four weeks (Unsupervised Phase).
  Subjects in the control group will play cognitive oriented video games using Wii Big Brain Academy Degree program. BigBrain™ is a video gaming system which has games and exercises to improve cognitive function(identify, memorize, analyze, compute, and visualize). Subjects use the Wii handheld remote to participate in the games by pointing and clicking the remote to select on-screen answers in response to on-screen questions.
  Interventions: Device: Wii Big Brain Academy Degree program
- WiiNWALK Intervention (Experimental): The intervention group will also receive 40 minute supervised group training three times per week for a period of four weeks. Interventions conducted over the first week will be held at the clinic, while the remaining three weeks be conducted at the subject's home and supervised by the Trainer remotely. At the end of the four-week Supervised Phase, subjects will retain the Wii units and they will be encouraged to use the program on their own for an additional period of four weeks (Unsupervised Phase).
  The WiiNWALK protocol consists of performing Nintendo WiiFit activities. Subjects stand on the WiiFit balance board and interact with the WiiFit games through weight shifting or by using the Wii handheld remote control. The intervention protocol will include selected exercises consisting of: 1) Yoga 2) Balance Tasks 3) Strength training and 4) Aerobics.
  At the in-clinic sessions in Vancouver, a motion-sensing device will also record video and skeleton data of the participant.
  Interventions: Device: Nintendo Wii

INTERVENTIONS:
Device: Nintendo Wii — Subjects will receive the intervention for 40-minute sessions, 3x/week for 4 weeks. The interventions will be administered in combination of onsite group training and individualized home-based training.
  Arms: WiiNWALK Intervention
Device: Wii Big Brain Academy Degree program — Subjects will receive the intervention for 40-minute sessions, 3x/week for 4 weeks. The interventions will be administered in combination of onsite group training and individualized home-based training.
  Arms: Cognitive Games

SUMMARY:
WiiNWALK is a 4 week physical activity, with the intervention of a WiiFit, targeted to improve walking capacity in individuals with either a unilateral below-knee or above-knee amputation. This is a randomized control trial to evaluate the effectiveness of the WiiNWALK program in older (50+ years) community living adults with lower limb amputations (LLA).

Hypothesis: We expect the WiiNWALK intervention will have a treatment effect with improvement in functional walking capacity, compared to the control group who will only be playing cognitive games. Secondarily, a functional walking capacity will also include an improvement in lower extremity strength and balance, inter-limb gait symmetry, balance confidence along with participation in daily and social activities, locomotor capabilities and an increase in physical activities.

DETAILED DESCRIPTION:
Lower limb amputation (LLA) is prevalent among older Canadians. Estimates from 2003 suggest that > 2 million individuals were living with LLA in North America with an annual estimated 150,000 incident cases. Over 50% of these procedures are considered major, with 28% of individuals having a transtibial (TT) or below knee amputation and 26% having a transfemoral (TF) or above knee amputation. The WiiNWalk is designed to evaluate whether this intervention does improve the walking capacity of older adults through a series of balancing and other physical activities using the Wii balance board.

An improved walking capacity (ie: being able to walk a longer distance) may effect balance, strength, and fitness components that are critical to improve prosthetic walking. The ability to walk a longer distance may effect a person's lifestyle as it allows the individual to move around his/her environment independently which in turn impacts ones choice of daily and social activities and participation, and therefore providing them with more mobility, freedom and choice.

This study focuses on older adults because, according to Canadian Institute of Health Information data, 50-74 year old were 17 times more likely to have a LLA and individuals aged ≥ 75 were 36 times more likely to have a LLA.The primary reason for this exponential age-related increased incidence is the late stage effects of chronic diseases such as diabetes and vascular disease that are common in older adults.

If as anticipated, the WiiFit proves to increase walking capacity, it will provide a low cost method for those with LLA to have an accessible system that, due to the weight-shifting, balance and aerobic training nature of the Wii games, will serve as a therapeutic agent for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be at least 50 years of age and have a unilateral TT or TF amputation
* Use their prosthesis for at least two hours per day for the past 6 months
* Be cognitively able to engage in the program
* Have a television that will enable connection to Nintendo hardware

Exclusion Criteria:

* Are unable to communicate in English
* Cannot provide informed consent
* Have important medical conditions
* Have prosthetic fit issues (ie: pain and discomfort)
* Are currently enrolled in another formal exercise or training program

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
2 Minute Walk to assess walking speed and endurance improvement | Baseline, Post Intervention (1 month after baseline), 3 week Follow-Up
  Starting from a standing position, subjects are asked to walk as far as they can in a safe manner for two minutes over a flat out and back 80-metre course. The distance travelled to the nearest metre is recorded.
Change in Two Minute Walk Test from baseline | Post-Intervention (1 month from Baseline)
  To assess changes in the participant's walking speed and endurance, they will start from a standing position, subjects are asked to walk as far as they can in a safe manner for two minutes over a flat out and back 80-metre course. The distance traveled to the nearest meter is recorded.
Change in two minute walk test from 1 month assessment | Follow-Up (3 weeks from post-intervention)
  Starting from a standing position, subjects are asked to walk as far as they can in a safe manner for two minutes over a flat out and back 80-metre course. The distance travelled to the nearest metre is recorded.

SECONDARY OUTCOMES:
Physical Activity Scale for the Elderly (PASE) | Baseline, Post Intervention (1 month after baseline), 3 week Follow-Up
  The Physical Activity Scale for the Elderly (PASE) is a self-report measure that captures information on the frequency, duration, and intensity of various physical activities. The 10 item PASE is generally partitioned into two parts. Part one, Leisure Time Activity, has six items that capture information about individual's involvement in daily activities such as participating in light exercise during the past seven days. The response options are never, seldom, sometimes, or often. Information on the type and the average time spent engaging in the activity per day is also captured.
  Part two, Household Activity, has three yes/no items which ask about participation in daily activities such as dusting or washing dishes over the past week. The last question asks about involvement in paid or volunteer work over the past week. The PASE also asks about the number of hours per week as well as the amount of physical activity involved for the job or volunteer work.
Short Physical Performance Battery (SPPB) ability | Baseline
  Short Physical Performance Battery (SPPB) will be used to measure subjects' lower extremity function by scoring their ability to perform four tasks: double-leg standing balance (feet together, semi-tandem, tandem), single-leg standing balance, gait speed over 4 meters, and lower extremity strength (5x chair stands). Each task is scored from 0 (poor) to 4 (excellent). A total score will be generated by adding up the scores for individual tasks. We will look at overall and balance component scores.
Change in Physical Activity Scale of the Elderly (PASE) | Post-Intervention (1 month from baseline)
  The Physical Activity Scale for the Elderly (PASE) is a self-report measure that captures information on the frequency, duration, and intensity of various physical activities. The 10 item PASE is generally partitioned into two parts. Part one, Leisure Time Activity, has six items that capture information about individual's involvement in daily activities such as participating in light exercise during the past seven days. The response options are never, seldom, sometimes, or often. Information on the type and the average time spent engaging in the activity per day is also captured.
  Part two, Household Activity, has three yes/no items which ask about participation in daily activities such as dusting or washing dishes over the past week. The last question asks about involvement in paid or volunteer work over the past week. The PASE also asks about the number of hours per week as well as the amount of physical activity involved for the job or volunteer work.
Change in Physical Activity Scale for the Elderly (PASE) | Follow-Up (3 weeks from post-intervention)
  The Physical Activity Scale for the Elderly (PASE) is a self-report measure that captures information on the frequency, duration, and intensity of various physical activities. The 10 item PASE is generally partitioned into two parts. Part one, Leisure Time Activity, has six items that capture information about individual's involvement in daily activities such as participating in light exercise during the past seven days. The response options are never, seldom, sometimes, or often. Information on the type and the average time spent engaging in the activity per day is also captured.
  Part two, Household Activity, has three yes/no items which ask about participation in daily activities such as dusting or washing dishes over the past week. The last question asks about involvement in paid or volunteer work over the past week. The PASE also asks about the number of hours per week as well as the amount of physical activity involved for the job or volunteer work.
Change in Short Physical Performance Battery (SPPB) | Post Intervention (1 month from baseline)
  Short Physical Performance Battery (SPPB) will be used to measure subjects' lower extremity function by scoring their ability to perform four tasks: double-leg standing balance (feet together, semi-tandem, tandem), single-leg standing balance, gait speed over 4 meters, and lower extremity strength (5x chair stands). Each task is scored from 0 (poor) to 4 (excellent). A total score will be generated by adding up the scores for individual tasks. We will look at overall and balance component scores.
Change in Short Physical Performance Battery from Post-Intervention | Follow-Up (3 weeks from post intervention)
  Short Physical Performance Battery (SPPB) will be used to measure subjects' lower extremity function by scoring their ability to perform four tasks: double-leg standing balance (feet together, semi-tandem, tandem), single-leg standing balance, gait speed over 4 meters, and lower extremity strength (5x chair stands). Each task is scored from 0 (poor) to 4 (excellent). A total score will be generated by adding up the scores for individual tasks. We will look at overall and balance component scores.
Four Square Step Test (FSST) | Baseline, Post Intervention (1 month after baseline), 3 week Follow-Up
  The Four Square Step Test (FSST) will measure dynamic standing balance. Four canes are placed on the floor to create 4 squares. The subject will step in each square as fast as possible and with use of his/her walking aid if needed. At the end of the test, the subject would have moved forward, backward, left and right while stepping over low objects. It also involves multiple transfer of weight between feet while changing direction. This test is timed and faster times indicate better dynamic standing balance.

OTHER OUTCOMES:
Life Space Assessment (LSA) | Baseline
  The Life Space Assessment is a five-item questionnaire that will be used to measure the size of the spatial area that subjects move in their daily life, as well as the frequency of their mobility within a certain time frame.
StepwatchTM Activity Monitor (SAM) | Baseline
  Activity Monitor (SAM) will be mounted on the ankle of prosthetic limb to monitor and record information regarding the number of steps per time interval to indicate the amount of physical activity performed in the community.
Health Utility Index (HUI3) | Baseline
  The HUI3 is a brief questionnaire that asks subjects about their health status.
Walking While Talking Test | Baseline
  Subjects walk flat 20 feet (six metres) on a flat course, turn around, and walk 20 feet back to the start while reciting the letters of the alphabet (a, b, c, ...) aloud. They repeat this routine while reciting alternate letters of the alphabet (a, c, e, …) aloud. Subjects will be asked to pay attention to both walking and talking. The difference in time (to the nearest second) to complete the simple and complex walks is calculated with higher differences suggesting poorer ability to cope with dual tasks (e.g., greater need to focus on walking).
Locomotor Capabilities Index in Amputees | Baseline
  This is composed of 14 items that ask questions about subject's ability to perform different locomotor activities with their prosthesis on. Items are scored on a 5-level ordinal scale from 0 (not able) to 4 (able to accomplish the activity alone without ambulation aids). The total score ranges from 0 to 56, with higher scores indicating greater locomotor capabilities with the prosthesis and less dependence on assistance.
Fall Calendar | Baseline
  This will be used to document the number of falls, circumstances (eg: cause, location, assistive device used or not) and consequences subject have had (eg/ medical visit, injury) over the course of study.
Change in Life Space Assessment from Baseline | Post Intervention (1 month from Baseline)
  The Life Space Assessment is a five-item questionnaire that will be used to measure the size of the spatial area that subjects move in their daily life, as well as the frequency of their mobility within a certain time frame.
Change in Life Space Assessment from Post Intervention | Follow-Up (3 weeks from Post-Intervention)
  The Life Space Assessment is a five-item questionnaire that will be used to measure the size of the spatial area that subjects move in their daily life, as well as the frequency of their mobility within a certain time frame.
Change in Fall calendar from Baseline | Post-Intervention (1 months from Baseline), Follow-Up (3 weeks from Post-Intervention), 62 weeks
  This will be used to document the number of falls, circumstances (eg: cause, location, assistive device used or not) and consequences subject have had (eg/ medical visit, injury) over the course of study.
Change in Health Utility Index (HUI3)from baseline | Post-Intervention (1 month from baseline)
  The HUI3 is a brief questionnaire that asks subjects about their health status.
Change in Health Utility Index (HUI3) | Follow-Up (3 weeks from Post-Intervention)
  The HUI3 is a brief questionnaire that asks subjects about their health status.
Change in Locomotor Capabilities Index in Amputees from Baseline | Post-Intervention (one month from baseline)
  This is composed of 14 items that ask questions about subject's ability to perform different locomotor activities with their prosthesis on. Items are scored on a 5-level ordinal scale from 0 (not able) to 4 (able to accomplish the activity alone without ambulation aids). The total score ranges from 0 to 56, with higher scores indicating greater locomotor capabilities with the prosthesis and less dependence on assistance.
Change in Locomotor Capabilities Index in Amputees from Post-Intervention | Follow-Up (3 weeks from Post-Intervention)
  This is composed of 14 items that ask questions about subject's ability to perform different locomotor activities with their prosthesis on. Items are scored on a 5-level ordinal scale from 0 (not able) to 4 (able to accomplish the activity alone without ambulation aids). The total score ranges from 0 to 56, with higher scores indicating greater locomotor capabilities with the prosthesis and less dependence on assistance.
Change in Walking While Talking Test from baseline | Post-Intervention (1 month from baseline)
  Subjects walk flat 20 feet (six metres) on a flat course, turn around, and walk 20 feet back to the start while reciting the letters of the alphabet (a, b, c, ...) aloud. They repeat this routine while reciting alternate letters of the alphabet (a, c, e, …) aloud. Subjects will be asked to pay attention to both walking and talking. The difference in time (to the nearest second) to complete the simple and complex walks is calculated with higher differences suggesting poorer ability to cope with dual tasks (e.g., greater need to focus on walking).
Change in Walking While Talking test from Post-intervention | Follow-Up (3 weeks from Post-intervention)
  Subjects walk flat 20 feet (six metres) on a flat course, turn around, and walk 20 feet back to the start while reciting the letters of the alphabet (a, b, c, ...) aloud. They repeat this routine while reciting alternate letters of the alphabet (a, c, e, …) aloud. Subjects will be asked to pay attention to both walking and talking. The difference in time (to the nearest second) to complete the simple and complex walks is calculated with higher differences suggesting poorer ability to cope with dual tasks (e.g., greater need to focus on walking).
Qualitative Interviews | 1 month post-intervention
  We will be conducting optional qualitative interviews with participants from the Vancouver site. The purpose of the qualitative interviews is to learn more about their personal experiences using either the brain or physical activity video game-based training programs.

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - Glenrose Rehabilitation Centre, Edmonton, Alberta
  - Holy Family Hospital, Vancouver, British Columbia
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Parkwood Hospital, London, Ontario

REFERENCES:
- [Derived] Tao G, Miller WC, Eng JJ, Esfandiari E, Imam B, Lindstrom H, Payne MW. Group-based telerehabilitation intervention using Wii Fit to improve walking in older adults with lower limb amputation (WiiNWalk): A randomized control trial. Clin Rehabil. 2022 Mar;36(3):331-341. doi: 10.1177/02692155211061222. Epub 2021 Nov 29. PMID 34841917
- [Derived] Imam B, Miller WC, Finlayson HC, Eng JJ, Payne MW, Jarus T, Goldsmith CH, Mitchell IM. A Telehealth Intervention Using Nintendo Wii Fit Balance Boards and iPads to Improve Walking in Older Adults With Lower Limb Amputation (Wii.n.Walk): Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2014 Dec 22;3(4):e80. doi: 10.2196/resprot.4031. PMID 25533902